CLINICAL TRIAL: NCT04719819
Title: Spinal Anaesthesia for Caesarean Section: Descriptive Multicentre Study
Acronym: CesAR
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2020 BONNIN
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia, Spinal; Nonemergency Cesarean Section
Keywords: Anaesthesia, Spinal; Caesarean Section; Hyperbaric bupivacaine; Hemodynamic management after spinal anaesthesia; Maternal experience
MeSH Terms: interventions — Anesthesia, Spinal; Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Usual pratice: Assessment of usual practices
  Interventions: Procedure: Spinal anaesthesia for caesarean section

INTERVENTIONS:
Procedure: Spinal anaesthesia for caesarean section — Descriptive questionnaire with open and closed questions, to be completed during the procedure

SUMMARY:
Most of caesarean sections can be performed under spinal anaesthesia. Its major advantages are reliability and fast onset. However, dose of hyperbaric bupivacaine used, combination with adjuvants, hemodynamic management, and impact of these measures on maternal experience are not uniform. This study aims to describe practices of spinal anaesthesia for caesarean section in France to improve practices, guide new studies and establish protocols.

DETAILED DESCRIPTION:
Most of caesarean sections can be performed under spinal anaesthesia. Its major advantages are reliability and fast onset. However, techniques of spinal anaesthesia are varied. Dose of hyperbaric bupivacaine used may shifted, varying intensity of sensor block but also hemodynamic side effect. Likewise, use of adjuvant is frequent and differs between centres. Management of the maternal hemodynamic is also discussed. While it is recognized that intraoperatively vascular filling alone is not effective, use of vasopressors is not unequivocal. For example, recent studies support the use of norepinephrine.

Finally, maternal experience is a hot topic. Although insufficient anaesthesia is rare, it is often overlooked. There are few recommendations on the intraoperative treatment of insufficient anaesthesia and to the management of post-traumatic stress that it lead to.

The objective of this study is to describe practices of spinal anaesthesia for scheduled or non-emergency caesarean section (also named "green code") in France by detailing several points:

Technique of spinal anaesthesia:

* The anaesthesia solution used (doses and adjuvants)
* Management of hemodynamic
* Management of insufficient anaesthesia
* Maternal experience It aims to make an inventory of practices, to orient future studies, guide practice and the realization of protocols.

It is an observational study unfolds from 2021 to 2022. It concerns 11 French centres and 600 women. Data are collected with an online questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Affiliation to social security system
* Scheduled or elective Caesarean section (green code) under spinal anesthesia

Exclusion Criteria:

* Refusal to participate in the study
* Code red Caesarean section or general anesthesia decision
* Complicated" Caesarean section or combined spinal-epidural technique
* Presence of an epidural catheter
* Performing a combined spinal-epidural technique (even if the epidural catheter is not used)
* Contraindication to spinal anaesthesia (coagulation disorder, vertebral-medullary pathologies)
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy
Study Population: Women with spinal anaesthesia scheduled or non-emergency caesarean section
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Maternal data | Day of surgery
  Ad hoc Questionnaire
Obstetrical data | Day of surgery
  Ad hoc Questionnaire
Spinal procedure | Day of surgery
  Ad hoc Questionnaire
Haemodynamic management | Day of surgery
  Ad hoc Questionnaire
Maternal experience | Day of surgery
  Ad hoc Questionnaire

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CHU, Clermont-Ferrand
  - CHU, Grenoble
  - Hôpital Emile Roux, Le Puy-en-Velay
  - CHU, Lille
  - HCL, Lyon
  - CHU, Nancy
  - CHU, Nîmes
  - APHP Cochin, Paris
  - APHP Necker, Paris
  - APHP Trousseau, Paris
  - Hôpital Jacques Puel, Rodez